CLINICAL TRIAL: NCT00981149
Title: Duloxetine for Treatment of Painful Temporomandibular Joint Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00040504
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- duloxetine study drug (Experimental): Drug
  Interventions: Drug: duloxetine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: duloxetine — Evaluate the analgesic effect of 30 mg duloxetine twice daily in comparison to matching placebo at baseline (BL) and follow up over a six week period
  Other Names: Cymbalta
  Arms: duloxetine study drug
Drug: Placebo — Placebo match duloxetine for 6 week period.
  Arms: Placebo

SUMMARY:
Temporomandibular joint disorders (TMJD) are a family of musculoskeletal disorders that represent the most common chronic orofacial pain condition. TMJD is associated with persistent pain in the region of the temporomandibular joint and muscles of the head and neck. The purpose of this study is to test duloxetine (Cymbalta) as a potential treatment for chronic facial pain. Duloxetine is FDA approved as an antidepressant and for the chronic pain conditions of fibromyalgia and diabetic neuropathy. Chronic facial pain may be linked to Temporomandibular Joint Disorder (TMJD) which currently has no standard treatment.

DETAILED DESCRIPTION:
The proposed clinical trial will evaluate the analgesic and adverse effects of duloxetine, a serotonin and norepinephrine reuptake inhibitor, in comparison to placebo in patients with temporomandibular joint disorder (TMJD). Duloxetine is approved as an antidepressant and has been shown effective in the chronic pain conditions of fibromyalgia and diabetic neuropathy. Decrease in pain and dysfunction and improvement in quality of life and global satisfaction will be assessed over 6 weeks. Successful demonstration of a therapeutic effect may provide a basis for clinical use of duloxetine in patients with painful TMJD.

Background

TMJD is a heterogeneous family of musculoskeletal disorders associated with the temporomandibular joint, the periauricular region, and the muscles of the head and neck. TMJD has been identified as a major cause of nondental, chronic pain in the craniofacial region, second only to headache (NIH Technology Assessment Conference, 1997). Although few population-based epidemiological studies have been conducted, studies report the prevalence of TMJD as up to 20% in the adult population (Dworkin et al 1990, Schiffman et al 1990). Dworkin and colleagues conducted a series of studies of TMJD using valid and reliable examination and survey procedures (Von Korff et al 1988, Dworkin et al 1990, Carlsson and LeResche 1995) and identified 12.1% of the test population with painful TMJD with a female to male ratio of approximately 7:1. They also found the annual incidence of developing TMJD to be just over 2% with females tending to show a higher incidence rate than males (Von Korff et al 1993). Hence, TMJD is common in the general population, but it has also been reported that about 20% of patients with early signs and symptoms of TMJD will progress to a persistent pain state (Schiffman et al 1990).

Several studies of TMJD suggest that patients exhibit a state of CNS hypersensitivity similar to that reported in fibromyalgia (Maixner et al 1995, Maixner et al 1998, Sarlani and Greenspan 2003, Sarlani et al 2004) that contributes to the predicted widespread characteristics of the pain. Genetic factors that impact increased pain sensitivity, psychological traits and sex differences, and often coupled with environmental stress, may result in a phenotype that is vulnerable to musculoskeletal disease and susceptible to selective pharmacological treatment.

In addition to female gender, two other factors predict an elevated incidence of these disorders: a history of musculoskeletal pain at other body sites and quality of life symptoms typically associated with depression (Von Korff et al 1988, Raphael and Marbach 2001, John et al 2003). Patients diagnosed with fibromyalgia often exhibit concurrent orofacial symptomatology that mimics TMJD (Ta et al 2002, Sarlani and Greenspan 2003, Sarlani et al 2004). These observations and findings suggest that drugs useful for depression, affecting musculoskeletal systems, and effective in improving central monoaminergic neurotransmission, are prime candidates for the treatment of TMJD. For these reasons, we hypothesize that selective noradrenergic or combined noradrenergic and serotonin reuptake inhibitors should be effective for TMJD.

Lack of research has resulted in a paucity of evidence-based treatment approaches for TMJD (Antczak- Bouckoms 1995, List 2003). While NSAIDs are sometimes used, there is little evidence for their effectiveness for TMJD (Dionne 1997, Gordon et al 1990, 1991) except in frank joint involvement (Ta et al 2004), and gastrointestinal and renal toxicity limit their long-term use (Gabriel et al 1991, Allison et al 1992, Schafer et al 1995, Champion et al 1997) for treatment of chronic pain. Use of opioids has been discouraged for this chronic pain condition due to the limitations of long-term use for this drug class (DeNucci et al 1996, Dionne 1997). The most promising pharmacologic therapy for TMJD to date has been antidepressants, but it is important to note that indication for their clinical use has primarily been extrapolated from other chronic pain conditions (McQuay et al 1992, Onghena et al 1992). Only two randomized controlled trials have examined one of the tricyclic antidepressants (amitryptyline) for TMJD specifically (Sharav et all 1987, Rizzatti-Barbosa 2003). Amitryptyline for TMJD demonstrated an average response rate of 40% in these two studies, but its adverse effects result in a large percentage of patients discontinuing the drug before achieving pain relief (DeNucci et al 1996), resulting in an unfavorable risk to benefit ratio (Zitman et al 1990). Taken together, there has been insufficient evidence to adopt a pharmacologic standard of care for treatment of TMJD.

Duloxetine has shown efficacy for several chronic pain conditions (Sultan 2008) including fibromyalgia, and appears to be more effective in women than men (Arnold 2004, 2005). It is well tolerated and effective at a dose of 60 mg daily ( Sultan 2008). Studies in patients with fibromyalgia (Arnold 2004, 2005), diabetic neuropathy (Goldstein 2005), low back pain (Skijaravala 2008), and osteoarthritis (Chappell 2008) have shown an analgesic effect at this dose with fewer adverse effects and a lower drop out rate than higher doses. In the proposed study, subjects randomized to the intervention will use 60 mg of duloxetine given as 30 mg twice daily after a one-week period of 30 mg daily.

Given the prevalence of TMJD and the controversial nature of non-pharmacologic therapies such as occlusal alteration, intraoral devices, and surgery, the need exists for pharmacologic treatment that is efficacious but avoids adverse effects that discourage long-term use. This study will also provide a basis for future investigations of the etiology and management of painful TMJD.

Purpose/Objective of this study? TMJD represents a prototypic musculoskeletal disease whose characteristics of associated depression, comorbidity of fibromyalgia, female prevalence, increased CNS sensitivity to pain, and likely genetic differences among susceptible individuals, makes it a disorder that will likely be responsive to duloxetine treatment.The overall objective is to investigate duloxetine as a potential treatment for chronic pain of TMJD. We hypothesize that subjects receiving duloxetine will experience greater analgesia than those receiving placebo.

Specifically we will:

1. Evaluate the analgesic effect of 30 mg duloxetine twice daily in comparison to matching placebo at baseline (BL) and follow up over a six week period using the primary outcome measure of change in spontaneous pain. 2. Evaluate jaw functioning and evoked pain as measured by range of motion, pain with jaw movement, and pain pressure thresholds. 3. Assess frequency of adverse effects and their impact on patient global satisfaction and study adherence. 4. Examine sleep in relationship to pain. 5. Evaluate genetic susceptibilty to pain and response to duloxetine.

These aims and outcome measures are listed in prioritized order. The study is powered on the primary outcome measure of spontaneous pain; other measures are exploratory. The study is not powered to detect subgroup differences for variables such as gender, depression, type of TMJD diagnosis, or concurrent medications, as described later in the Analysis Plan.

Research Design: The study is a double blind, placebo-controlled parallel groups prospective study of duloxetine versus placebo. Subjects will be randomized to the investigational treatment group (duloxetine) or the placebo group. At the time of enrollment they will be randomly assigned to study drug or placebo by block randomization for order in a 1:1 ratio. Subjects will be provided acetominophen as a rescue analgesic to use if they feel their pain is not adequately controlled. The examiners and subjects will be blind to the group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic TMJD pain of two weeks duration
* Age 18 and older
* Confirmed craniofacial pain of nonodontogenic origin by the Research Diagnostic Criteria for temporomandibular disorders (TMD-RDC)
* Concomitant medications are permitted, except those which may convey analgesia
* Females who are neither pregnant, as verified by a urine-based pregnancy test, nor breast-feeding
* Female subjects of childbearing potential and those who are post-menopausal for less than 2 years must be using/willing to use a medically approved method of contraception (i.e., oral, transdermal or implanted contraceptive devices, intrauterine device, diaphragm, condom, abstinence, or surgical sterility during the course of the study
* Able to read and comprehend the rating scales, study instructions, and the consent form
* Pain score of 4 or greater on the baseline VAS (0-10)

Exclusion Criteria:

* Undergone any type of TMJ surgery or had TMJ growth disturbances, neoplasm, or injury to the TMJ area within the past six months
* Taking analgesic or anti-inflammatory drugs, steroids, antidepressants, antiepileptics, or opioid medications that may confound the assessment of analgesia
* Subjects with primary psychiatric diagnosis of major depression, suicidal ideation, or history of suicide attempt as assessed by medical history and the Mini International Neuropsychiatric Interview (MINI) are not eligible. Subjects with a score above average or higher in comparison with normative scores on the Beck Depression Inventory (BDI) will be allowed to participate
* Exclusions based on the effects of duloxetine:

  * Known hypersensitivity to duloxetine or its inactive ingredients
  * Subjects with: renal impairment or end stage renal disease; urinary retention or hesitation, delayed gastric emptying; substantial alcohol use or evidence of chronic liver disease, hepatic insufficiency and hepatotoxicity; bleeding disorders, orthostatic hypotension, uncontrolled high blood pressure; recent history of myocardial infarction or unstable coronary artery disease; seizure disorder, history of bipolar disorder or mania, general anxiety disorder (GAD); hyponatremia; uncontrolled narrow-angle glaucoma.
  * Treatment with an monoamine oxidase inhibitor (MAOI) within 30 days of randomization, or potential need to use an MAOI during the study or within 5 days of discontinuation of the drug
  * Concomitant use of medications such as: NSAIDs, warfarin, aspirin or other drugs that affect coagulation; Thioridazine and inhibitors of CYP1A2 which affect metabolism of duloxetine; serotonergic drugs like triptans and MAOIs which increase the risk of Serotonin Syndrome; drugs that affect gastric acidity
* Contraindications to acetaminophen use
* Ever been treated with duloxetine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Gordon, DDS MPH, PhD, Principal Investigator — University of Maryland Dental School
Locations (1):
- University of Maryland Dental School, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine Study Drug | Placebo
Started | 12 | 12
Completed | 10 | 9
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine Study Drug | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Customized [Count of Participants; unit: Participants]
  18 to 65 years | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 4 | 12
  Black | 4 | 6 | 10
  Hispanic | 0 | 1 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Pain as Measured by Visual Analog Scale at Baseline and at End of 6 Weeks.
Description: Measurements from zero to 100 with 100 being the worst pain by Visual Analog Scale (VAS).
Time Frame: 1, 3, 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine Study Drug | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale
  1 week | 42.9 (14.5) | 51.4 (19)
  3 weeks | 30.4 (18) | 44 (25)
  6 weeks | 34.8 (23.7) | 36.7 (26)

2. Secondary Outcome: Evoked Pain Via Algometry .
Description: Assessment of evoked pain using digital palpation examination at 18 predefined bodily sites.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Pain pressure threshold (kg/cm2)
Arm/Group | Duloxetine Study Drug | Placebo
Number analyzed (Participants) | 12 | 12
Pain pressure threshold (kg/cm2) | 311.9 (115.8) | 300.8 (80.9)

ADVERSE EVENTS:
Time Frame: 1, 3, and 6 weeks
Arm/Group | Duloxetine Study Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duloxetine Study Drug (N=10) | Placebo (N=9)
Headache (General disorders) | 10 | 9
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 | 9
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No